CLINICAL TRIAL: NCT07284485
Title: A Phase 2 Trial of Nadunolimab for Current or Former Smokers With High-risk Lung Nodules.
Brief Title: Immunoprevention for High-risk Lung Lesions
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Robert Samstein (Other)
Collaborators: Cantargia AB (Industry)
Responsible Party: Sponsor-Investigator, Robert Samstein, Associate Professor, Icahn School of Medicine at Mount Sinai
Organization: Icahn School of Medicine at Mount Sinai (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: STUDY-25-00757; PRMC-25-050 (Other: Icahn School of Medicine at Mount Sinai)
Record Dates: First submitted 2025-12-08; First posted 2025-12-16 (Actual); Last update posted 2025-12-16 (Actual); Status verified 2025-12

CONDITIONS: High-risk Lung Nodules
Keywords: High-risk Lung nodules; Nadunolimab; immunoprevention; tobacco smokers 20 pack-years; multi-focal part-solid nodules; immunomodulatory compounds

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Nadunolimab (Experimental): 10mg/kg Nadunolimab administered every 3 weeks for 4 doses
  Interventions: Biological: Nadunolimab

INTERVENTIONS:
Biological: Nadunolimab — Nadunolimab will be administered 10mg/kg intravenously every 3 weeks for 4 doses

SUMMARY:
The main purpose of this study is to assess nadunolimab as an immunoprevention strategy for high-risk lung nodules in participants who are current or former tobacco smokers. The study may last up to 5 years for each participant.

DETAILED DESCRIPTION:
The trial is a single-arm phase 2 of trial nadunolimab as an immunoprevention strategy for high-risk lung nodules. Eligible patients include patients who currently smoke or have previously smoked more than 20 pack-years and have high-risk lung nodules. High-risk nodules are defined as multifocal part-solid nodules (> or equal to 2 lesions, at least one with solid component <9mm) with evidence of progression on at least one annual follow-up CT scan.

The trial will be run as a Simon's optimal two-stage design, with an initial enrollment of 20 patients in the first stage. If only one patient shows response in stage 1 the arm will be stopped for futility. And if at least two patients have a documented regression of at least one high-risk part solid nodule, without significant DLT, then prior to opening Simon's Two Stage expansion slots the researchers will submit an amendment to the FDA with updated toxicity data regarding the first 20 patients enrolled. The researchers will await FDA approval of this amendment before the researchers would start enrollment of the additional patients beyond the first 20 patients. If FDA approves then an additional 36 patients will be enrolled in stage 2. From the complete arm of 56 patients if 5 or more patients achieve a response then nadunolimab will be declared efficacious. and a larger phase 2-3 trial could be developed to more formally test the efficacy of the drug. As such, statistical comparisons will still be compared to the historical control which represents the current standard treatment of observation. The researchers anticipate accrual to take up to 2 years from the time of initiation resulting an accrual of 1-3 patient per month. The researchers expect to replace up to 5% of the patients. Hence, the total number of patients that should be enrolled to obtain the aforementioned 56 evaluable patients is 59 if study is expanded to stage 2.

ELIGIBILITY:
Inclusion Criteria:

* Participants must be current or former tobacco smokers (>20 pack years)
* Participants must have multi-focal part-solid nodules (>2 lesions, at least one with solid component <9mm) with evidence of progression on at least one annual follow-up CT scan.
* Participants must not meet criteria for surgical intervention at the time of enrollment.
* Patient must be willing and able to provide blood samples (12 green-top tubes, roughly 100mL) at the five time points indicated in the Study Calendar.
* Age ≥ 18 years.
* ECOG 0-1. The exception will be Participants carrying long term disability (such as cerebral palsy) where the disability is not acute nor progressive, and unlikely to significantly affect their response to therapy. This must be documented in screening clinic visit note by investigator.
* Women of child-bearing potential and men must agree to use adequate contraception prior to study entry, for the duration of study participation, and for 1 month and 6 months following completion of therapy, for woman and men, respectively. Should a woman become pregnant or suspect she is pregnant while participating in this study, she should inform her treating physician immediately. A female of child-bearing potential is any woman (regardless of sexual orientation, having undergone a tubal ligation, or remaining celibate by choice) who meets the following criteria:

  * Has not undergone a hysterectomy or bilateral oophorectomy; or
  * Has not been naturally postmenopausal for at least 24 consecutive months
* Ability to understand and the willingness to sign a written informed consent.
* Adequate organ and marrow function as defined below:

  * Hematologic
  * - Absolute neutrophil count (ANC) ≥1,500 /mcL
  * - Platelets ≥100,000 /mcL
  * - Hemoglobin ≥9 g/dL
  * Renal*
  * - Serum creatinine ≤1.5 X upper limit of normal (ULN) OR Measured or calculated (calculated per institutional standard) creatinine clearance (GFR can also be used in place of creatinine or CrCl) ≥60 mL/min GFR for patient with creatinine levels > 1.5 X institutional ULN
  * Hepatic*
  * - Serum total bilirubin ≤ 1.5 X ULN OR Direct bilirubin ≤ ULN for
  * - Participants with total bilirubin levels > 1.5 ULN
  * - AST or ALT ≤ 2.5 X ULN
  * - Albumin >2.5 mg/dL

    * If laboratory criteria are not met due to what the investigator determines to be a biologic cause (e.g. Gilbert's syndrome causing elevated bilirubin or excessive muscle mass affecting creatinine) or drug-related cause (e.g. elevating in transaminases due to HAART therapy, elevated INR due to anticoagulation) then the specific lab values will not be used to exclude patient from this trial. This determination will be made by PI.

Exclusion Criteria:

* Any pulmonary nodule with a solid component >8mm.
* Patients may not be receiving any other investigational agents at the time of enrollment.
* Uncontrolled intercurrent illness prior to starting therapy including, but not limited to, ongoing or active infection requiring antibiotics (exception is a brief (≤10days) course of antibiotics to be completed before initiation of treatment), symptomatic congestive heart failure, unstable angina pectoris, or psychiatric illness/social situations that would limit compliance with study requirements.
* Patients must not be pregnant or nursing due to the potential for congenital abnormalities and the potential of this regimen to harm nursing infants.
* Has a diagnosis of immunodeficiency or is receiving systemic steroid therapy or any other form of immunosuppressive therapy within 7 days prior to the first dose of trial treatment. Exception: Patients on chronic steroids (more than 4 weeks at stable dose) equivalent to ≤ 10mg prednisone will not be excluded.
* Has active autoimmune disease that has required systemic treatment in the past 1 year (i.e. with use of disease modifying agents, corticosteroids or immunosuppressive drugs). Exception: Replacement therapy (e.g. thyroxine, insulin, or physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency, etc.) is acceptable.
* Has a history or current evidence of any condition, therapy, or laboratory abnormality that might confound the results of the trial, interfere with the patient's participation for the full duration of the trial, or is not in the best interest of the patient to participate, in the opinion of the treating Investigator.
* Known HIV positive with detectable viral load, or anyone not on stable anti-viral (HAART) regimen, or with <200 CD4+ T cells/microliter in the peripheral blood. HIV testing is not required for patients with no known history of HIV.
* Has known Hepatitis B or active Hepatitis C (e.g., HCV RNA [qualitative] is detected). HBV and HCV testing is not required for patients with no known history of these viruses.
* History of allogeneic hematopoietic cell transplantation or solid organ transplantation.
* Receipt of a live vaccine, etanercept, or tumor necrosis factor-alpha inhibitors within 30 days of planned start of study drug
* Documented allergic or hypersensitivity response to any protein therapeutics (e.g., recombinant proteins, vaccines, intravenous immune globulins, monoclonal antibodies, receptor traps)Principal investigator believes that for one or multiple reasons the patient will be unable to comply with all study visits, or if they believe the trial is not clinically in the best interest of the patient.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 59 (Estimated)
Dates: Start 2025-12-15 (Estimated); Primary Completion 2027-12-15 (Estimated); Study Completion 2029-12-17 (Estimated)

PRIMARY OUTCOMES:
Response rate | 3 months from initiation of study drug
  Response rate is defined as the proportion of patients who achieve this regression on imaging obtained at 3 months. Regression will be defined as ≥20% reduction in the largest diameter of at least one lung nodule at 3 months after initiation of biologic therapy.

SECONDARY OUTCOMES:
Number of adverse events | 6 months from initiation of study drug.
  The safety and tolerability of nadunolimab will be assessed according to the NCI Common Toxicity Criteria for Adverse Events (CTCAE), version 5.0.
Number of participants with regression of nodules | 2 years from initiation of study drug.
  The regression of nodules defined as ≥20% reduction in the largest diameter of at least one lung nodule at 3 months after initiation of biologic therapy., at subsequent follow-up imaging timepoints past 3 months for up to 2 years
Progression-free survival | From treatment initiation until progression of disease, initiation of anti-cancer therapy or death, up to 2 years, whichever comes first.
  Progression-free survival based on the time from treatment initiation until the time of radiographic evidence of progression of disease, initiation of anti-cancer therapy or death, whichever comes first

CONTACTS AND LOCATIONS:
Overall Officials: Robert M Samstein, MD, PhD, Principal Investigator — Icahn School of Medicine at Mount Sinai; Thomas Marron, MD, PhD, Study Chair — Icahn School of Medicine at Mount Sinai
Locations (1):
- Icahn School of Medicine at Mount Sinai, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No
The completed dataset is the sole property of the Sponsor-Investigator's institution and should not be exported to third parties, except for authorized representatives of appropriate Health/Regulatory Authorities, without permission from the Sponsor-investigator and their institution.

REFERENCES:
- [Background] LaMarche NM, Hegde S, Park MD, Maier BB, Troncoso L, Le Berichel J, Hamon P, Belabed M, Mattiuz R, Hennequin C, Chin T, Reid AM, Reyes-Torres I, Nemeth E, Zhang R, Olson OC, Doroshow DB, Rohs NC, Gomez JE, Veluswamy R, Hall N, Venturini N, Ginhoux F, Liu Z, Buckup M, Figueiredo I, Roudko V, Miyake K, Karasuyama H, Gonzalez-Kozlova E, Gnjatic S, Passegue E, Kim-Schulze S, Brown BD, Hirsch FR, Kim BS, Marron TU, Merad M. An IL-4 signalling axis in bone marrow drives pro-tumorigenic myelopoiesis. Nature. 2024 Jan;625(7993):166-174. doi: 10.1038/s41586-023-06797-9. Epub 2023 Dec 6. PMID 38057662
- [Background] Becker D, Stana J, Prendes C, Ali A, Pichlmaier M, Peterss S, Tsilimparis N. The Use of Short Dilator Tip in Endovascular Branched Arch Repair: A Case Series. J Endovasc Ther. 2024 Oct 18:15266028241283713. doi: 10.1177/15266028241283713. Online ahead of print. PMID 39422219
- [Background] Ridker PM, MacFadyen JG, Thuren T, Everett BM, Libby P, Glynn RJ; CANTOS Trial Group. Effect of interleukin-1beta inhibition with canakinumab on incident lung cancer in patients with atherosclerosis: exploratory results from a randomised, double-blind, placebo-controlled trial. Lancet. 2017 Oct 21;390(10105):1833-1842. doi: 10.1016/S0140-6736(17)32247-X. Epub 2017 Aug 27. PMID 28855077
- [Background] Garon EB, Lu S, Goto Y, De Marchi P, Paz-Ares L, Spigel DR, Thomas M, Yang JC, Ardizzoni A, Barlesi F, Orlov S, Yoshioka H, Mountzios G, Khanna S, Bossen C, Carbini M, Turri S, Myers A, Cho BC. Canakinumab as Adjuvant Therapy in Patients With Completely Resected Non-Small-Cell Lung Cancer: Results From the CANOPY-A Double-Blind, Randomized Clinical Trial. J Clin Oncol. 2024 Jan 10;42(2):180-191. doi: 10.1200/JCO.23.00910. Epub 2023 Oct 3. PMID 37788412
- [Background] Tan DSW, Felip E, de Castro G, Solomon BJ, Greystoke A, Cho BC, Cobo M, Kim TM, Ganguly S, Carcereny E, Paz-Ares L, Bennouna J, Garassino MC, Schenker M, Kim SW, Brase JC, Bury-Maynard D, Passos VQ, Deudon S, Dharan B, Song Y, Caparica R, Johnson BE. Canakinumab Versus Placebo in Combination With First-Line Pembrolizumab Plus Chemotherapy for Advanced Non-Small-Cell Lung Cancer: Results From the CANOPY-1 Trial. J Clin Oncol. 2024 Jan 10;42(2):192-204. doi: 10.1200/JCO.23.00980. Epub 2023 Dec 1. PMID 38039427
- [Background] International Early Lung Cancer Action Program Investigators; Henschke CI, Yankelevitz DF, Libby DM, Pasmantier MW, Smith JP, Miettinen OS. Survival of patients with stage I lung cancer detected on CT screening. N Engl J Med. 2006 Oct 26;355(17):1763-71. doi: 10.1056/NEJMoa060476. PMID 17065637
- [Background] Henschke CI, Yip R, Sun Q, Li P, Kaufman A, Samstein R, Connery C, Kohman L, Lee P, Tannous H, Yankelevitz DF, Taioli E, Rosenzweig K, Flores RM; I-ELCAP; IELCART Investigators. Prospective Cohort Study to Compare Long-Term Lung Cancer-Specific and All-Cause Survival of Clinical Early Stage (T1a-b; </=20 mm) NSCLC Treated by Stereotactic Body Radiation Therapy and Surgery. J Thorac Oncol. 2024 Mar;19(3):476-490. doi: 10.1016/j.jtho.2023.10.002. Epub 2023 Oct 6. PMID 37806384
- [Background] Garlanda C, Dinarello CA, Mantovani A. The interleukin-1 family: back to the future. Immunity. 2013 Dec 12;39(6):1003-18. doi: 10.1016/j.immuni.2013.11.010. PMID 24332029
- [Background] Nemoto H, Honjo M, Okamoto M, Sugimoto K, Aihara M. Potential Mechanisms of Intraocular Pressure Reduction by Micropulse Transscleral Cyclophotocoagulation in Rabbit Eyes. Invest Ophthalmol Vis Sci. 2022 Jun 1;63(6):3. doi: 10.1167/iovs.63.6.3. PMID 35653121
- [Background] Baas P, Scherpereel A, Nowak AK, Fujimoto N, Peters S, Tsao AS, Mansfield AS, Popat S, Jahan T, Antonia S, Oulkhouir Y, Bautista Y, Cornelissen R, Greillier L, Grossi F, Kowalski D, Rodriguez-Cid J, Aanur P, Oukessou A, Baudelet C, Zalcman G. First-line nivolumab plus ipilimumab in unresectable malignant pleural mesothelioma (CheckMate 743): a multicentre, randomised, open-label, phase 3 trial. Lancet. 2021 Jan 30;397(10272):375-386. doi: 10.1016/S0140-6736(20)32714-8. Epub 2021 Jan 21. PMID 33485464
- [Background] Focker J, Huang L, Caling AL, Fischer M, Ihle A, Hodgson T, Kattner F. Enhanced auditory serial recall of recently presented auditory digits following auditory distractor presentation in blind individuals. Q J Exp Psychol (Hove). 2024 Dec 16:17470218241300115. doi: 10.1177/17470218241300115. Online ahead of print. PMID 39501663
- [Background] Krammer F. A correlate of protection for SARS-CoV-2 vaccines is urgently needed. Nat Med. 2021 Jul;27(7):1147-1148. doi: 10.1038/s41591-021-01432-4. No abstract available. PMID 34239135